CLINICAL TRIAL: NCT05225259
Title: Expanded Access of LOXO-260 in Participants With RET Mutant or RET Fusion Tumors Refractory to Prior RET Selective TKI Treatment
Brief Title: Expanded Access for LOXO-260 in Participants With Cancer Caused by an Abnormal RET Gene That Did Not Respond/is no Longer Responding to Treatment With a Type of Drug Called a RET Inhibitor
Status: No longer available | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LOXO-260 Expanded Access
Record Dates: First submitted 2022-01-28; First posted 2022-02-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms
Keywords: Solid tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: LOXO-260 — Oral
  Other Names: LY3838915

SUMMARY:
Expanded access for participants with cancer caused by an abnormal RET gene that did not respond/is no longer responding to treatment with a type of drug called a RET inhibitor.

The treating physician/investigator contacts Loxo Oncology, Inc. when, based on their medical opinion, a patient meets the criteria for expanded access.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer with RET mutant (medullary thyroid cancer [MTC] or multiple endocrine neoplasia type 2 [MEN2] tumors) or RET fusion (solid tumors) advanced/metastatic tumors that have become refractory to RET selective tyrosine kinase inhibitor (TKI) treatment, who are not eligible or able to participate in an ongoing LOXO-260 clinical trial and are medically suitable for treatment with LOXO-260.
* Patients tumor must have developed RET solvent front mutations (eg G810X) after RET selective treatment.
* Have progressed or are intolerant to standard therapy, or no standard therapy option exists, or in the opinion of the investigator, are unlikely to derive significant clinical benefit from standard therapy
* Have adequate organ function
* Patients must reside in a country where the LOXO-NGR-21001 study (NCT05241834) is not open or recruiting.

Exclusion Criteria:

* Currently enrolled in an ongoing clinical study of LOXO-260 or another second generation RET inhibitor
* Clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to study treatment; ongoing cardiomyopathy; or current prolongation of the QT interval corrected for heart rate using Fridericia's formula (QTcF) interval greater than 470 milliseconds
* Clinically significant malabsorption syndrome
* Pregnant or lactating
* Eastern Cooperative Oncology Group (ECOG) performance status 3 or 4
* Patients harboring known activating bypass alterations outside RET (eg. EGFR, ALK, RAS etc) that may confer resistance to LOXO-260

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Emin Avsar, MD, Study Director — Loxo Oncology, Inc.